CLINICAL TRIAL: NCT05290675
Title: Impact of Sample Type and Assay Time on the Performance of the Quantra QPlus System
Brief Title: Quantra QPlus Sample Type Comparison
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-042
Record Dates: First submitted 2022-01-13; First posted 2022-03-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Coagulation Defect; Bleeding
Keywords: Cardiac surgery; Quantra; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Quantra QPlus System — Whole blood coagulation testing system

SUMMARY:
This is a single center prospective observational study to compare QPlus parameter measurements in arterial and venous blood samples collected in parallel from patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
In this single center prospective observational study, 40 cardiac surgery subjects will enrolled, each with parallel artrial and venous samples collected at 3 time points to yield 120 matched samples for analysis on the Quantra System with the QPlus Cartridge.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for cardiac surgery, utilizing cardiopulmonary bypass, or including placement of a ventricular assist device
* Subject is ≥18 years
* Subject or subject's legally authorized representative is willing to participate and he/she has signed a consent formr.

Exclusion Criteria:

* Subject is younger than 18 years
* Subject is pregnant
* Subject is incarcerated at the time of the study
* Subject is affected by a condition that, in the opinion of the surgical team, may pose additional risks
* Subject, or subject's legally aurthorized representative is able to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Comparison of QPlus Clot time (CT) in arterial and venous samples | During cardiac surgery
  Coagulation function assessed in two sample types
Comparison of QPlus Clot time with Heparinase (CTH) in arterial and venous samples | During cardiac surgery
  Coagulation function assessed in two sample types
Comparison of Clot stiffness (CS) determined with Quantra QPlus Cartridge in arterial and venous samples | During cardiac surgery
  Measure of the overall shear modulus or strength/quality of the clot determined using SEER sonorheometry assessed in two sample types
Comparison of QPlus Platelet Contribution to Clot stiffness (PCS) in arterial and venous samples | During cardiac surgery
  Measure of the shear modulus or strength/quality of the clot contributed by platelets determined using SEER sonorheometry assessed in two sample types
Comparison of QPlus Fibrinogen Contribution to Clot stiffness (FCS) in arterial and venous samples | During cardiac surgery
  Measure of the shear modulus or strength/quality of the clot contributed by fibrinogen determined using SEER sonorheometry assessed in two sample types

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No